CLINICAL TRIAL: NCT06982300
Title: Towards Improved Therapy Selection and Targeted Treatment for Nasopharyngeal Carcinoma: a Proof-of-concept Pilot Study for Somatostatin Receptor 2 Imaging With [68Ga]Ga-DOTA-TOC PET/CT.
Brief Title: SSTR2 Imaging With [68Ga]Ga-DOTA-TOC PET/CT in NPC
Acronym: NACASOR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21477; 2025-520689-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-25; First posted 2025-05-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]Ga-DOTA-TOC PET imaging (Experimental)
  Interventions: Other: [68Ga]Ga-DOTA-TOC PET imaging

INTERVENTIONS:
Other: [68Ga]Ga-DOTA-TOC PET imaging — Patients will undergo [68Ga]Ga-DOTA-TOC PET imaging before and 3 weeks after start of standard of care treatment with induction chemotherapy or CRT, unless the baseline scan shows no tracer uptake in the tumor, in that case the scan will not be repeated.
  Patients will receive 120 MBq [68Ga]Ga-DOTA-TOC intravenously and will be scanned up to 20 minutes, 60 minutes after tracer injection, after acquisition of a low dose CT for attenuation correction.
  The investigators will use archival tissue of the diagnostic biopsy for SSTR2 staining. If there is not sufficient tumor tissue available, a new biopsy will be performed after the baseline PET scan.
  Blood samples will be drawn before the start, during and after finishing therapy at 3 or 4 different time points, depending on the treatment schedule.

SUMMARY:
This is an investigator-initiated, single-center clinical trial designed to evaluate the feasibility of [68Ga]Ga-DOTA-TOC positron emission tomography (PET) scan in patients with Epstein-Barr virus (EBV) related nasopharyngeal carcinome (NPC) prior to and three weeks after the start of induction chemotherapy or concurrent chemoradiotherapy (CRT). Archival tumor tissue from the diagnostic biopsy will be used to perform somatostatin receptor 2 (SSTR2) immunohistochemistry (IHC). Blood samples will be drawn at baseline, after three weeks, after completion of induction chemotherapy if applicable, and after CRT.

ELIGIBILITY:
Inclusion Criteria:

* Stage IB-IVA NPC (AJCC 9th edition), EBV positive determined by Epstein-Barr virus-encoded RNA (EBER).
* Planned treatment with induction chemotherapy or CRT without induction chemotherapy.
* Age ≥ 18 years.
* Signed informed consent.
* Willingness and ability to comply with all protocol required procedures.
* Negative serum pregnancy test at screening in women of childbearing potential.
* Archival tumor tissue available or consent to undergo a tumor biopsy procedure.

Exclusion Criteria:

* Previous treatment with chemotherapy or radiotherapy for NPC.
* Treatment with any investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to [68Ga]Ga-DOTA-TOC injection.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or that may affect the interpretation of the results or render the patient at high risk from complications.
* Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Inability to lie in supine position for 25 minutes.
* Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of assessing tumor SSTR2 expression | From the day of the first study scan within one week before the start of treatment to the day of the second study scan three weeks after the start of treatment
  Determine feasibility of assessing tumor SSTR2 expression in patients with EBV-associated NPC in a non-endemic region by repeat [68Ga]Ga-DOTA-TOC PET imaging.

SECONDARY OUTCOMES:
[68Ga]Ga-DOTA-TOC uptake in the primary tumor and lymph node metastase | From the day of the first study scan within one week before the start of treatment to the day of the second study scan three weeks after the start of treatment
  Determine [68Ga]Ga-DOTA-TOC uptake in the primary tumor and lymph node metastases in patients with EBV-related NPC, at baseline and early after the start of curative intent treatment, consisting of CRT with or without induction chemotherapy.
[68Ga]Ga-DOTA-TOC distribution | From the day of the first study scan within one week before the start of treatment to the day of the second study scan three weeks after the start of treatment
  Normal tissue and organ distribution of [68Ga]Ga-DOTA-TOC in NPC patients defined by standard uptake value (SUV)
Comparison [68Ga]Ga-DOTA-TOC uptake with SSTR expression | The day of the first study scan within one week before the start of treatment
  Comparison of tumor [68Ga]Ga-DOTA-TOC uptake on the baseline study PET scan with SSTR2 expression on the tumor biopsy, determined by IHC.

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje F. Oosting, MD, PhD, Principal Investigator — University Medical Center Groningen, Dept. of Medical Oncology, Hanzeplein 1, 9713 GZ Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The decision whether or not to share IPD will be made after consultation of the PI.